CLINICAL TRIAL: NCT06611748
Title: Evaluation of a Simple Neuroprosthesis for Restoration of Hand Function in Cervical Spinal Cord Injury
Brief Title: Restoration of Hand Function in Cervical SCI
Acronym: KeyGrip
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Megan Moynahan, Principal Investigator, MetroHealth Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00000625; ID573-FY24-25 (Other Grant/Funding Number: Ohio Department of Education)
Record Dates: First submitted 2024-09-18; First posted 2024-09-25 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2024-11

CONDITIONS: Spinal Cord Injury Cervical
Keywords: Cervical Spinal Cord Injury (SCI)

STUDY DESIGN:
Intervention Model Description: KeyGrip is an implantable peripheral nerve stimulator that is being studied for its ability to provide coordinated activation of innervated paralyzed muscles. KeyGrip will be configured to activate nerves of the upper extremity (arm and hand) in order to facilitate movements such as hand opening and/or closing. The study will evaluate participants; grasp strength and ability to manipulate standard objects with each participant serving as their own control, comparing stimulation ON vs. OFF.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- KeyGrip device implantation (Experimental): The KeyGrip system components will be implanted in a single surgical procedure, lasting up to 90 minutes.
  For this study, a small receiver will be placed under the skin in the forearm. Up to four stimulating electrodes(investigational) will be surgically placed in muscles of the hand or arm. Wires from these electrodes will be tunneled beneath the skin and connected to the receiver device located in the forearm.
  The study participant will control the electrical stimulation by using a phone app that communicates to a power unit that is placed on the skin over the receiver. Following implantation of the device, periodic evaluations will be performed to assess their condition, and the operation and usefulness of the device.
  Depending on the study participant's usage level, they may need to recharge the batteries every night.
  Interventions: Device: Key Grip; Device: Implanted Key Grip Electrodes

INTERVENTIONS:
Device: Key Grip — KeyGrip is an implantable peripheral nerve stimulator that is being studied for its ability to provide coordinated activation of innervated paralyzed muscles. KeyGrip will be configured to activate nerves of the upper extremity (arm and hand) in order to facilitate movements such as hand opening and/or closing
Device: Implanted Key Grip Electrodes — The KeyGrip System uses modified implanted wires (called "electrodes") that deliver stimulation to the muscles. These electrodes are also investigational.

SUMMARY:
The purpose of this study is to evaluate a new method of restoring hand function to people with spinal cord injury. Current methods to restore hand function include tendon transfers and nerve transfers. This study will evaluate the grasp strength that can be achieved with a small, implantable stimulator.

KeyGrip is an investigational device that works by activating paralyzed muscles with low levels of electrical current. The word "investigational" means the study device is still being tested in research studies and is not approved by the U.S. Food and Drug Administration (FDA) for the use being studied.

Hypothesis. The study is designed to explore the feasibility of this approach; no hypothesis is planned at this stage

DETAILED DESCRIPTION:
The purpose of this study is to evaluate an alternative method of restoring hand function to people with spinal cord injury. Current methods to restore hand function include tendon transfers (surgery that moves working muscles and tendon to replace a nonworking muscle and tendon) and nerve transfers (surgery that reroutes a healthy nerve to connect to a damaged nerve and restore function or sensation). This study will evaluate the grasp strength and ability to manipulate objects that can be achieved with a small (2 inches long) implantable stimulator. The device we are using to achieve this is the Nalu Medical Peripheral Nerve Stimulator.

Nalu Medical Peripheral Nerve Stimulator is a stimulator currently used to treat chronic pain. The Nalu Medical Peripheral Nerve Stimulator is currently cleared for marketing by the U.S. Food and Drug Administration (FDA) for the use of spinal cord stimulation and peripheral nerve stimulation to block pain signals. The Nalu Medical Peripheral Nerve Stimulator has not been approved by the FDA for the use being tested in this study. We intend to use this device to activate paralyzed muscles. When being used for the purpose of this study, we will refer to the device as the KeyGrip System.

The KeyGrip System is an investigational use of an FDA approved device (The Nalu Medical Peripheral Nerve Stimulator) that works by activating paralyzed muscles with low levels of electrical current. The word "investigational" means the way we are using the device is still being tested in research studies and is not approved by the (FDA) for the use being studied. This study will use the KeyGrip System to try to restore hand function to people with spinal cord injury.

What is involved in this study?

If the participant chooses to be in this study, the participant will undergo the following procedures:

* a screening procedure that involves using surface electrical stimulation (that is, stimulation using pads placed on the skin) to evaluate whether the participants muscles can be activated with electrical stimulation.
* Following this, the participant will undergo an evaluation of their current hand grasp strength, and the ability to perform a test of hand grasp that involves manipulating standard objects.
* If the participants are a candidate for the study, participants will undergo surgery to implant the KeyGrip system, after which the hand and forearm will be immobilized in a cast for 3 weeks to protect the electrodes from movement.
* Participants will then have the implant programmed to provide grasp and will be trained in how to use the system to perform activities.
* Participants will then be able to use the system at home for exercise and for functional activities.
* Over the course of the first year, participants will return at 3-, 6-, and 12-months to evaluate grasp strength, and ability to manipulate standard objects.
* It is important to note that investigators do not plan to remove the study device after participation in the study ends. If participants wish to remove the study device after finishing participating or if participants withdraw from the study, a surgery to remove the device can be scheduled.

Participants will be in this research study for one year, after which participants may continue to use the device. Participants will continue to be contacted by the research team to monitor any adverse events participants may experience.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults 18 years of age or older;
* Cervical spinal cord injury as defined by: a) International Standard for Neurological Classification of Spinal Cord Injury motor level of C1 through C7; and b) American Spinal Injury Association Impairment Scale (AIS) grade A, B, or C;
* Six months or more post-injury (neurostability);
* Neurologically stable following any nerve transfers affecting the upper extremity (typically, one-year post-surgery);
* Musculoskeletally and neurologically stable following any tendon transfers affecting the upper extremity (typically 6 months post-surgery).
* Peripheral nerve innervation to upper extremity muscles, including Grade 3/5 or higher Stimulated Manual Muscle Testin at least two of the muscles in one arm:
* Good proximal voluntary upper extremity strength as defined by biceps/ brachialis / brachioradialis strength of 2/5 or higher on Manual Muscle Testing the side intended for implantation;
* Medically stable; and
* Able to understand and provide informed consent;

Exclusion Criteria:

* Other neurological conditions (Multiple Sclerosis, diabetes with peripheral nerve involvement);
* Associated peripheral nerve / brachial plexus injury;
* Progressive Spinal Cord Injury;
* Active implantable medical device (AIMD) such as a pacemaker or defibrillator;
* Active untreated infection such as urinary tract infection or pneumonia;
* Active pressure injury;
* History of coagulopathy, HIV, cardiopulmonary disease, bradycardia, poorly controlled autonomic dysreflexia, or chronic obstructive pulmonary disease that would preclude safe participation in the trial as determined by the investigator;
* Unhealed fractures that prevent functional use of arm;
* Extensive upper extremity denervation (fewer than two excitable hand muscles);
* Involvement in other ongoing clinical studies that exclude concurrent involvement in this study;
* Currently pregnant (neuroprosthesis implantation delayed until no longer pregnant based on self-report); Urine or serum testing will happen during the pre-surgery evaluation.
* Presence of disease that might interfere with participant safety, compliance, or evaluation of the condition under study;
* Other significant medical findings that, in the opinion of the investigator, preclude safe participation in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Grasp-Release Test (GRT) | baseline, 3-weeks post treatment, 12-weeks post treatment, 26-week post treatment, 52 weeks post treatment
  The GRT is a standardized pick-and-place test that evaluates two prehensile patterns (palmar and lateral grasp) using standardized objects of different weights and sizes that are designed to mimic objects encountered in daily life.

SECONDARY OUTCOMES:
Grasp Strength | baseline, 3 weeks post treatment, 12 weeks post treatment, 26-week post treatment, 52 weeks post treatment
  Lateral grasp strength is measured with and without the stimulation to identify changes in force that contribute to object acquisition and task performance
  Palmer Lateral grasp strength is measured with and without the stimulation to identify changes in force that contribute to object acquisition and task performance.
Activities of Daily Living Abilities Test | baseline, 12-weeks post treatment, 26-weeks post treatment, and 52-weeks post treatment
  Functional goals will be identified by the participant. Participants will be evaluated in their level of independence in performing the tasks both with and without stimulation. Participants will rate the task on a scale of +(better), 0(same), - worse after they complete each task with the device on verse with the device off.
  This test allows us to measure the impact of the device on the participants individual functional goals.
Canadian Occupational Performance Measure (COPM) | baseline, 12-weeks post treatment, 26-weeks post treatment, and 52-weeks post treatment
  The COPM is a client-centered assessment that measures a participant's perceived level of activity performance and satisfaction with that performance. The participant identifies the goals / activities and performance is assessed with and without the neuroprosthesis.
  Importance is rated on a 10-point scale with 1=not important at all and 10=extremely important Performance is rated on 10-point scale with 1=not able to do it at all and 10=able to do it extremely well Satisfaction is rated on a 10-point scale with 1=not satisfied and 10=extremely satisfied
  Change in importance, performance and satisfaction is calculated over time. Higher score is better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Moynahan, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: KeyGrip website — https://www.keygrip.co/